CLINICAL TRIAL: NCT01581372
Title: A Community Based Approach to Dyslipidemia Management: Pharmacist Prescribing to Achieve Cholesterol Targets (RxACT Study)
Brief Title: A Community Based Approach to Dyslipidemia Management: Pharmacist Prescribing to Achieve Cholesterol Targets
Acronym: RxACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Ross T. Tsuyuki, Director and Professor of Medicine, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020054
Record Dates: First submitted 2012-03-05; First posted 2012-04-20 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist care (Experimental)
  Interventions: Other: Pharmacist care
- Usual care (No Intervention)

INTERVENTIONS:
Other: Pharmacist care — Pharmacist prescribing, education, drug management
  Arms: Pharmacist care

SUMMARY:
Background:

Cardiovascular disease (CVD) is the cause of one-third of all deaths in Canada. One important risk factor for CVD is dyslipidemia. The Canadian Health Measures survey, which was conducted from 2007-2009, found that roughly 36% of Canadians had unhealthy levels of LDL. Despite strong evidence and clear practice guidelines for the management of this risk factor, it remains poorly treated.

Pharmacists are front-line primary care professionals who see patients at risk for cardiovascular disease more frequently than other healthcare professionals. As such, pharmacists have the opportunity to systematically and proactively identify patients with undertreated dyslipidemia, as one public health approach to chronic disease management.

The objective of this study is to evaluate the effect of enhanced pharmacist care (i.e., participant identification, assessment, care plan development, education/counseling, prescribing/titration of lipid-lowering medications and close follow-up) on the proportion of participants achieving target LDL-cholesterol levels.

Hypothesis: Enhanced pharmacist care will result in a more significant decrease in LDL-c levels, than that observed in the usual care patients.

Design:

This is a randomized controlled trial of enhanced pharmacist care. The study will be conducted in twelve community pharmacies in Alberta, including several Safeway Pharmacies. The participant population will be composed of adults with uncontrolled dyslipidemia as defined by the 2009 Canadian Dyslipidemia Guidelines. The primary intervention will be pharmacist directed dyslipidemia care. Participants randomized to usual care will receive usual care from their pharmacist and physician.

Study Implications:

To the investigators knowledge, this study is the first randomized trial of pharmacist prescribing in dyslipidemia. This study will have important implications for improving patients' access to care, especially as most provinces are proceeding with granting additional prescribing authority to pharmacists. The ability to conduct this study in a province where pharmacists already have the ability to prescribe is unique. The results will also encourage more pharmacists to get involved in cardiovascular prevention and will increase the number of prescribers in the area of dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* All adults >18 years of age
* Suboptimal dyslipidemia control, defined as:
* high risk (coronary disease (stroke/TIA), cerebrovascular disease, peripheral arterial disease, diabetes, or Framingham Risk Score >20%) and LDL-c >2.0 mmol/L
* moderate risk (Framingham Risk Score 10-19%) and LDL-c >3.5 mmol/L
* moderate risk (Framingham risk score 10-19%) in males >50 years or females >60 years with an LDL-c of ≤3.5 mmol/L and hs-CRP > 2.0 mg/L (measured twice 1-2 weeks apart)

Exclusion Criteria:

* Participant unwilling to use statins,
* Participant has a demonstrated intolerance to statins,
* Participant is pregnant or nursing
* Participant has renal impairment (defined as a creatinine ≤30 mL/min) or hepatic dysfunction
* Participant is unwilling or unable to attend follow-up visits, or is unlikely to adhere to study procedures (due to cognitive limitations, severe psychiatric disorders or alcoholism)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving their target LDL-c in the intervention versus usual care group | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ross T Tsuyuki, PharmD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Safeway, Calgary, Alberta
  - London Drugs, Lethbridge, Alberta